CLINICAL TRIAL: NCT04949477
Title: Intranasal Dexmedetomidine Versus Oral Paracetamol as a Pre-anaesthetic Medication in Pediatric Age Group Undergoing Adenotonsillectomy: A Randomised Clinical Trial
Brief Title: Intranasal Dexmedetomidine Versus Oral Paracetamol as a Pre-anaesthetic Medication in Pediatric Age Group
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Fatma Ahmed Abdel Fatah, Lecturer, Benha University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8-5-2021
Record Dates: First submitted 2021-06-25; First posted 2021-07-02 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Anxiety
Keywords: Dexmedetomidine; Paracetamol; Preoperative anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Dexmedetomidine; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (D) (Active Comparator): The patient will receive intranasal dexmedetomidine.
  Interventions: Drug: Dexmedetomidine
- Group (P) (Active Comparator): The patient will receive paracetamol orally.
  Interventions: Drug: paracetamol

INTERVENTIONS:
Drug: Dexmedetomidine — the patient will receive intranasal dexmedetomidine at a dose of 1 μg/kg to the patient 45 min. before the procedure.
  Other Names: precedex
  Arms: Group (D)
Drug: paracetamol — the patient will receive paracetamol orally [Rx paracetamol 250 mg/ml] at a dose of 20 mg/kg given to the patient 45 min before the procedure by drinking.
  Other Names: cetal
  Arms: Group (P)

SUMMARY:
Pre-operative anxiety is a major problem in children because it produces undesired results on induction and postoperative outcome. Dexmedetomidine is a highly specific alpha 2 adrenergic receptor agonist. Studies suggest that Dexmetomidine administration is safe as it is less invasive and have a short half-life.

Paracetamol is a potent physical pain killer. It also reduces psychological reactivity and blunts physical and social pain.

Adenotonsillectomy is one of the most common surgeries performed in pediatric age groups, so it is important to reduce pre-operative anxiety in those children.

DETAILED DESCRIPTION:
Pre-operative anxiety is a major problem in children because it produces undesired results on induction and postoperative outcome. Dexmedetomidine is a highly specific alpha 2 adrenergic receptor agonist. Studies suggest that Dexmetomidine administration is safe as it is less invasive and have a short half-life.

Paracetamol is a potent physical pain killer. It also reduces psychological reactivity and blunts physical and social pain.

Adenotonsillectomy is one of the most common surgeries performed in pediatric age groups, so it is important to reduce pre-operative anxiety in those children.

The objective of this descriptive study is to compare the efficacy of dexmedetomidine and paracetamol premedication, measuring the degree of anxiety in the children prepared for adenotonsillectomy when they are separated from their parents.

ELIGIBILITY:
Inclusion Criteria:

* The patients who are clinically free or with controlled medical condition [ASA I or ASA II].
* Age between 2 to 8 years.

Exclusion Criteria:

* ASA III or ASA IV.
* Age greater than 8 years.
* Parents' refusal to participate in the study.
* Patients with obstructive sleep apnea.
* Patients with known allergy or hypersensitivity reaction to any of the drugs used in the study.
* Patients with nasal infection or nasal pathology.

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 86 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Preoperative anxiety | After 50 minutes of drug administration.
  Modified Yale preoperative anxiety score (m-Yale PAS) before intravenous catheterization. In m-Yale PAS, anxiety was assessed based on their activities, (1-4) emotional expression, (1-4) Vocalization, (1-6) state of arousal (1-4) and interaction with family members.(1-4) The minimum of score is five (minimum anxiety) and the maximum is 22 which means severe anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Banha Faculity of Medicine, Banhā, Elqalyoubea, Egypt

IPD SHARING:
Plan to Share IPD: Undecided